CLINICAL TRIAL: NCT05597449
Title: Impact of YouTube Videos and Health Literacy on Postoperative Healthcare Utilization Following Pediatric Urologic Surgery
Brief Title: Surgical Patient Education in Pediatric Urology
Acronym: Uro Surg HL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Julie, Pediatric Urology acting instructor, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00003161
Record Dates: First submitted 2022-10-21; First posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Intervention Model Description: Families randomized by urologic surgery type to receive access to YouTube video link
Who Masked: Participant, Care Provider
Masking Description: Participants (caregivers) blinded to the intervention and outcomes and care providers blinded to the study group assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video group (Experimental): Access to YouTube videos and written postoperative instructions
  Interventions: Behavioral: YouTube videos on care after urologic surgery
- Control group (No Intervention): Access to written instructions only

INTERVENTIONS:
Behavioral: YouTube videos on care after urologic surgery — Supplemental educational videos regarding care following pediatric urologic surgery
  Arms: Video group

SUMMARY:
Randomized study to assess the impact of supplemental educational YouTube videos on postoperative healthcare utilization following ambulatory pediatric urologic surgery

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of patients age <18 years old undergoing ambulatory pediatric urologic surgery

Exclusion Criteria:

* Caregivers that decline participation

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Total number of episodes (Postoperative healthcare utilization) | 30 days following surgery
  Episodes of postoperative calls, messages, add-on clinic visits, Urgent Care or Emergency Department visits. Each caregiver-initiated call, message, or visit will count as an individual episode. Multiple calls, messages, and visits will each be counted toward a total number of episodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No